CLINICAL TRIAL: NCT03954873
Title: Glucagon-like Peptide 2 - a Glucose Dependent Glucagonotropic Hormone?
Acronym: GLANCE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Gentofte, Copenhagen (Other)
Responsible Party: Principal Investigator, Filip Krag Knop, Clinical Professor, University Hospital, Gentofte, Copenhagen
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: H-18046965
Record Dates: First submitted 2019-05-15; First posted 2019-05-17 (Actual); Last update posted 2020-11-04 (Actual); Status verified 2020-11

CONDITIONS: Glucose Metabolism Disorders; Endocrine or Metabolic Disease
Keywords: GLP-2; Glucagon
MeSH Terms: conditions — Glucose Metabolism Disorders; Metabolic Diseases | interventions — Glucagon-Like Peptide 2; Sodium Chloride; Glucose; Insulin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Hyperglycaemia + GLP-2 (Experimental): Glucose + GLP-2
  Interventions: Other: Glucagon-like peptide 2; Other: Glucose
- Hyperglycaemia + Placebo (Active Comparator): Glucose + saline
  Interventions: Other: Saline; Other: Glucose
- Hypoglycaemia + GLP-2 (Experimental): Insulin + glucose + GLP-2
  Interventions: Other: Glucagon-like peptide 2; Other: Glucose; Other: Insulin
- Hypoglycaemia + Saline (Active Comparator): Insulin + glucose
  Interventions: Other: Saline; Other: Glucose; Other: Insulin
- Euglycaemia + GLP-2 (Experimental): GLP-2
  Interventions: Other: Glucagon-like peptide 2
- Euglycaemia + Placebo (Active Comparator)
  Interventions: Other: Saline

INTERVENTIONS:
Other: Glucagon-like peptide 2 — Human glucagon-like peptide 2
  Arms: Euglycaemia + GLP-2; Hyperglycaemia + GLP-2; Hypoglycaemia + GLP-2
Other: Saline — Placebo
  Arms: Euglycaemia + Placebo; Hyperglycaemia + Placebo; Hypoglycaemia + Saline
Other: Glucose — 20% (w/v) glucose infusion for regulating plasma glucose
  Arms: Hyperglycaemia + GLP-2; Hyperglycaemia + Placebo; Hypoglycaemia + GLP-2; Hypoglycaemia + Saline
Other: Insulin — Actrapid (insulin) for lowering plasma glucose
  Arms: Hypoglycaemia + GLP-2; Hypoglycaemia + Saline

SUMMARY:
Infusion of glucagon-like peptide 2 (GLP-2) during euglycaemia, hypoglycaemia and hyperglycaemia and evaluation of the effect on glucagon secretion in healthy subjects.

DETAILED DESCRIPTION:
This is a cross-over, randomized, double-blinded study in which 10 participants will undergo 6 experimental days each. The participants will have their plasma glucose clamped at either euglycaemia (fasting level), hypoglycemia (2,5 mmol/l) or hyperglycemia (10 mmol/l) during infusion of GLP-2 or saline (placebo)

The six days will be as follows:

* Euglycaemia + Placebo
* Euglycaemia + GLP-2
* Hyperglycaemia + Placebo
* Hyperglycaemia + GLP-2
* Hypoglycaemia + Placebo
* Hypoglycaemia + GLP-2

The primary endpoint will be levels of plasma glucagon. Secondary endpoint will be levels of GLP-1, GLP-2, Insulin/C-peptide, OXM, Amino acids, CCK, Gastrin, norepinephrine, bile acids, FGF-19/FGF-21. Secondary endpoints will also include ultrasound scan of the gallbladder.

ELIGIBILITY:
Inclusion Criteria:

* Caucasian ethnicity
* Body mass index (BMI): 18.5-27 kg/m2
* Glycated haemoglobin (HbA1c) < 42 mmol/mol
* Normal haemoglobin (8.3-10.5 mmol/l)
* Informed and oral and written consent

Exclusion Criteria:

* Prediabetes, type 1 diabetes or type 2 diabetes or first-degree relatives with type 1 or type 2 diabetes
* Nephropathy (eGFR < 60 and/or albuminuria)
* Known liver disease and/or alanine transaminase (ALAT) or aspartate transaminase (ASAT) > 2 × upper normal limit
* Bilirubin > 25 μmol/l
* Known intestinal disease or previous surgery of the intestines
* Active or recent malignant disease
* Treatment with medicine that cannot be paused for 12 hours
* Any condition considered incompatible with participation by the investigators

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2019-01-31 (Actual); Primary Completion 2020-06-01 (Actual); Study Completion 2020-06-01 (Actual)

PRIMARY OUTCOMES:
Glucagon secretion | 110 minutes
  Assessed by difference in absolute plasma glucagon concentrations (measured in pmol/liter) and incremental (baseline-subtracted) area under curve (AUC) for plasma glucagon

SECONDARY OUTCOMES:
Plasma glucose | 110 minutes
  Measured in mmol/liter
GLP-1 | 110 minutes
  Glucagon-like peptide 1, Measured in pmol/liter
GLP-2 | 110 minutes
  Glucagon-like peptide 2, Measured in pmol/liter
Insulin | 110 minutes
  Measured in pmol/liter
GIP | 110 minutes
  Glucose dependent insulinotropic hormone, Measured in pmol/liter
OXM | 110 minutes
  Oxytomodulin, Measured in pmol/liter
Amino acids | 110 minutes
  Measured in pmol/liter
CCK | 110 minutes
  Cholecystokinin, Measured in pmol/liter
Gastrin | 110 minutes
  Measured in pmol/liter
FGF-19 | 110 minutes
  Fibroblast Growth factor 19, Measured in ng/mL
FGF-21 | 110 minutes
  Fibroblast Growth factor 21, Measured in ng/mL
Bile acids | 110 minutes
  Measured in nmol/ml
Norepinephrine | 110 minutes
  Measured in pmol/liter
GH | 110 minutes
  Growth hormone, Measured in nmol/ml
P1NP | 110 minutes
  Procollagen type I N-terminal propeptide (Bonemarker), Measured in nmol/ml
CTX | 110 minutes
  C-terminal telopeptide (Bonemarker), Measured in nmol/ml
Gallbladder ultrasound | 110 minutes
  Measuring of gallbladder size in respons to GLP-2
Glucose infusion | 90 minutes
  Amount of glucose infusion (20% v/w) in milliliters needed to clamp at isoglycemic levels (hyperglycemia and hypoglycemia) in respons to GLP-2
Blood pressure | 110 minutes
  Systolic (mmHg) and diastolic (mmHg) blood pressure in respons to GLP-2
Heart rate | 110 minutes
  Heart rate (beats/minutes) in respons to GLP-2
C-peptide | 110 minutes
  Measured in pmol/liter

CONTACTS AND LOCATIONS:
Overall Officials: Filip Krag Knop, MD, PhD, Study Director — Center for Clinical Metabolic Research
Locations (1):
- Center for Clinical Metabolic Research, Hellerup, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared with other researchers unless data management agreements are signed.